CLINICAL TRIAL: NCT07258407
Title: A Phase 1/2 Dose Escalation Trial With Administration Schedule Exploration Evaluating Single Agent TD001, a PSMA-Targeted Antibody-Drug Conjugate, in Patients With PSMA-Expressing Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Clinical Trial Evaluating the Safety of TD001 In Patients With PSMA-Expressing Metastatic Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: T.O.A.D. Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TD001-101; 2025-523273-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-Resistant Prostatic Cancer
Keywords: CRPC; PSMA; prostate-specific membrane antigen
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation design followed by RP2D cohort expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Sequential groups of participants receive TD001 at escalating doses
  Interventions: Drug: TD001
- RP2D dose expansion (Experimental): Groups of participants receive TD001 at the recommended Phase 2 doses (RP2Ds)
  Interventions: Drug: TD001

INTERVENTIONS:
Drug: TD001 — Intravenous (IV) infusion at protocol-defined doses and schedules until disease progression or other reason to end treatment

SUMMARY:
This study will evaluate the safety, tolerability, drug levels (pharmacokinetics) and preliminary antitumor activity of TD001, an antibody-drug conjugate (ADC) targeting prostate-specific membrane antigen (PSMA), in men with metastatic PSMA-expressing castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multicenter Phase 1/2 study with a dose escalation part to determine recommended Phase 2 doses (RP2Ds) of TD001 for further evaluation in an expansion part of the study. Multiple dosing schedules may be evaluated. The safety and preliminary efficacy endpoints of this study will support dose optimization in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient must fully understand the study requirements and voluntarily sign informed consent.
* PSMA-expressing metastatic CRPC with documented progression based on serum PSA, RECIST 1.1 with PCWG3, and/or bone disease.
* At least one measurable metastatic lesion per RECIST 1.1.
* Adequate organ function.
* Prior orchiectomy and/or ongoing androgen deprivation therapy.
* Prior treatment with at least one androgen receptor pathway inhibitor (ARPI) drug.

Exclusion Criteria:

* Previous treatment with strontium-89, samarium-153, rhenium-186, rhenium-188, radium-223, or hemi-body irradiation, within 6 months before treatment.
* Systemic anticancer therapy including an investigational agent within 28 days before treatment.
* Known hypersensitivity to the components of TD001, its analogs, or excipients.
* Current dyspnea at rest, other disease requiring continuous oxygen therapy, or history of pneumonitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (dose escalation) | Treatment + follow-up (estimated 9 months)
  Number of participants with dose-limiting toxicity; incidence of adverse events (AEs), serious AEs (SAEs), abnormal laboratory parameters, TD001 discontinuation or modification due to AEs, as assessed by CTCAE v6.0
Recommended Phase 2 doses (dose escalation) | Treatment + follow-up (estimated 9 months)
  Incidence of AEs, SAEs, abnormal laboratory parameters, TD001 discontinuation or modification due to AEs, as assessed by CTCAE v6.0
Safety/tolerability - incidence of AEs, SAEs, abnormal laboratory parameters (dose escalation + expansion) | Treatment + follow-up (estimated 21 months)
  AEs, SAEs, abnormal laboratory parameters by type, severity, and relatedness as assessed by CTCAE v6.0
Safety/tolerability - incidence of TD001 discontinuation or modification due to AEs (dose escalation + expansion) | Treatment + follow-up (estimated 21 months)
  AEs by type, severity, and relatedness as assessed by CTCAE v6.0

SECONDARY OUTCOMES:
Plasma PK - AUC | Estimated 6-8 months
  Area under the concentration-time curve for total ADC, total antibody, and unconjugated payload
Plasma PK - AUClast | Estimated 6-8 months
  Area under concentration-time curve from time zero to the last measurable concentration for total ADC, total antibody, and unconjugated payload
Plasma PK - AUCtau | Estimated 6-8 months
  Area under concentration-time curve from time zero to the end of the dosing interval for total ADC, total antibody, and unconjugated payload
Plasma PK - Cmax | Estimated 6-8 months
  Maximum concentration for total ADC, total antibody, and unconjugated payload
Plasma PK - Tmax | Estimated 6-8 months
  Time to maximum concentration for total ADC, total antibody, and unconjugated payload
Plasma PK - T1/2 | Estimated 6-8 months
  Terminal elimination half-life for total ADC, total antibody, and unconjugated payload
Plasma PK - Ctrough | Estimated 6-8 months
  Trough concentration for total ADC, total antibody, and unconjugated payload
PSA50 response rate | Treatment (estimated 8 months)
  ≥50% PSA decrease from baseline, per PCWG3
Overall response rate | Treatment (estimated 8 months)
  Best response of CR or PR per PCWG3-modified RECIST 1.1
PSA progression-free survival | Treatment + follow-up (estimated 21 months)
  Per PCWG3
Radiographic progression-free survival | Treatment + follow-up (estimated 21 months)
  per PCWG3-modified RECIST 1.1
Duration of response | Treatment + follow-up (estimated 21 months)
  For PSA and radiographic response
Disease control rate | Treatment (estimated 8 months)
  Best response of CR, PR or SD
Overall survival | Treatment + follow-up (estimated 21 months)
Immunogenicity - prevalance and incidence of ADAs | Treatment period + follow-up (estimated 9 months)
  ADAs against TD001 prior to first dose and at any time on treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No